CLINICAL TRIAL: NCT03499704
Title: A Multicenter, Randomized, Open-label, Two-arm, Phase 4 Study to Evaluate the Effect of Add-on Pioglitazone or Dapagliflozin in Subjects With Type 2 Diabetes Mellitus Inadequately Controlled by Dipeptidyl Peptidase-4 Inhibitor and Metformin Therapy
Brief Title: A Study to Evaluate the Effect of add-on Pioglitazone or Dapagliflozin in Participants With Type 2 Diabetes Mellitus Inadequately Controlled by DPP-4 Inhibitor and Metformin Therapy
Acronym: EPIDOTE
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Celltrion Pharm, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Alogliptin-Pio-4001; U1111-1207-8037 (Other: World Health Organization)
Record Dates: First submitted 2018-04-09; First posted 2018-04-17 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Drug therapy
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Pioglitazone; alogliptin; Metformin; dapagliflozin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pioglitazone + Alogliptin + Metformin (PAM) (Experimental): Pioglitazone 15 milligram (mg) and alogliptin 25 mg in fixed dose combination (FDC) tablet (SYR-322-4833), orally once daily and metformin greater than or equal to (>=) 500 mg, tablet, orally, twice a day for up to 26 weeks. At Week 12, if participants has HbA1c >=7.5%, pioglitazone dose will be titrated up to 30 mg based on investigator's opinion and up-titrated dose will be maintained up to Week 26.
  Interventions: Drug: Pioglitazone + Alogliptin; Drug: Metformin
- Dapagliflozin + Alogliptin + Metformin (DAM) (Active Comparator): Dapagliflozin 10 mg, tablet, orally, once daily with alogliptin 25 mg, tablet, orally, once daily, and metformin >=500 mg, tablet, orally, twice a day, for up to Week 26.
  Interventions: Drug: Alogliptin; Drug: Metformin; Drug: Dapagliflozin

INTERVENTIONS:
Drug: Pioglitazone + Alogliptin — Pioglitazone and Alogliptin FDC tablets
  Other Names: SYR-322-4833
  Arms: Pioglitazone + Alogliptin + Metformin (PAM)
Drug: Alogliptin — Alogliptin tablets.
  Arms: Dapagliflozin + Alogliptin + Metformin (DAM)
Drug: Metformin — Metformin tablets.
Drug: Dapagliflozin — Dapagliflozin tablets.
  Arms: Dapagliflozin + Alogliptin + Metformin (DAM)

SUMMARY:
The purpose of this study is to assess the pioglitazone plus alogliptin plus metformin is non-inferior to dapagliflozin plus alogliptin plus metformin on glycosylated haemoglobin (HbA1c) change from baseline at Week 26.

DETAILED DESCRIPTION:
The drug being tested in this study is Alogliptin Benzoate and Pioglitazone Hydrochloride FDC. This study will assess the efficacy of pioglitazone or dapagliflozin in participants with type 2 diabetes mellitus.

The study will enroll approximately 156 participants. Participants will be randomly assigned (by chance, like flipping a coin) to one of the two treatment groups.

* Pioglitazone 15 mg + Alogliptin 25 mg + Metformin >=500 mg
* Dapagliflozin 10 mg + Alogliptin 25 mg + Metformin >=500 mg

Based on investigators opinion at Week 12, if participant has HbA1c >=7.5%, dose of pioglitazone can be titrated up to 30 mg.

This multi-center trial will be conducted in Republic of Korea. The overall time to participate in this study is up to 36 weeks. Participants will make multiple visits to the clinic, and will be contacted by telephone 14 days after their last dose of drug for a follow-up assessment.

ELIGIBILITY:
Inclusion Criteria:

1. The subject is a regular outpatient with an has a historical diagnosis of type 2 diabetes.
2. The subject has metabolic syndrome as jointly defined by the International Diabetes Federation (IDF); National Heart, Lung, and Blood Institute (NHLBI) / American Heart Association (AHA); and International Association for the Study of Obesity (IASO). If any 3 of the following 5 risk factors are present, metabolic syndrome can be considered:

   * High waist circumference: male ≥ 90 cm, female ≥ 85 cm.
   * High TGs (drug treatment for high TGs is an alternate indicator): ≥ 150 mg/dL (1.7 mmol/L).
   * Low HDL-C (drug treatment for low HDL-C is an alternate indicator): < 40 mg/dL(1.0 mmol/L) in males, < 50 mg/dL (1.3 mmol/L) in females.
   * High blood pressure (antihypertensive drug treatment in a subject with a history of hypertension is an alternate indicator): Systolic ≥ 130 mmHg and/or diastolic ≥ 85 mmHg.
   * High fasting glucose (drug treatment of high glucose is an alternate indicator): ≥ 100 mg/dL.
3. The subject has been receiving a stable dose of DPP-4 inhibitor + metformin therapy with diet and exercise for ≥ 3 months prior to Randomization.
4. The subject has a HbA1c value between 7.0 and 11% inclusively within 28 days of Randomization via central laboratory test or after run-in period for 4 weeks via central laboratory test.

Exclusion Criteria:

1. The subject has type 1 diabetes, diabetic ketoacidosis, diabetic coma or diabetic precoma.
2. The subject has an active bladder cancer or a history of bladder cancer.
3. The use of any medications ie, oral or systemically injected glucocorticoids (including intra-articular injection), weight-loss drugs, insulin or other anti-diabetic drugs except DPP-4 inhibitor and metformin, within 3 months prior to randomization. Strong Cytochrome P450 2C8 (CYP2C8) inhibitors (eg, gemfibrozil, montelukast, quercetin, phenelzine) and CYP2C8 inducers (eg, rifampin) that in the opinion of the Investigator or Sponsor require treatment contraindicated during the study. The diuretics, angiotensin receptor blockers (ARBs), angiotensin-converting enzyme (ACE) -inhibitors and nonsteroidal anti-inflammatory drugs (NSAIDs) are to be used per product label with close monitoring under Investigator's supervision.
4. Has genetic problems such as galactose intolerance, Lapp lactose dehydrogenase deficiency or glucose-galactose uptake disorder, etc.
5. Has a history of alcohol abuse within 2 years prior to randomization.

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 133 (Actual)
Dates: Start 2020-02-11 (Actual); Primary Completion 2024-01-31 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Mean Change from Baseline in HbA1c at Week 26 | Baseline and Week 26

SECONDARY OUTCOMES:
Mean Change from Baseline in Homeostatic Model Assessment of Insulin Resistance (HOMA-IR) at Week 26 | Baseline and Week 26
  HOMA IR measures insulin resistance based on fasting glucose and insulin measurements: HOMA IR equal to (=) fasting insulin (micro unit per milliliter [mcU/mL])*fasting glucose (millimole per milliliter [mmol/mL])/22.5. A higher number indicates a greater insulin resistance.
Mean Change from Baseline in Serum Lipids at Week 26 | Baseline and Week 26
  The change from baseline in serum lipids (Total Cholesterol [TC], Low-density Lipoprotein Cholesterol [LDL-C], High-density Lipoprotein Cholesterol [HDL-C], Triglycerides [TGs]) will be analyzed using mixed model repeated measures (MMRM) model.
Number of Participants who Achieved an HbA1c Goal Target of Less than (<) 6.5 Percent (%) at Week 26 | Week 26

CONTACTS AND LOCATIONS:
Overall Officials: Medical Team, Study Director — Celltrionpharm Inc.
Locations (15):
- South Korea (15):
  - The Catholic University of Korea, Bucheon, St. Marys Hospital, Bucheon-si, Gyeonggi-do
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - The Catholic University of Korea, ST. Vincents Hospital, Suwon, Gyeonggi-do
  - Ajou University Hospital, Suwon, Gyeonggi-do
  - Inje University Haeundae Paik Hospital, Busan
  - Pusan National University Hospital, Busan
  - YeungNam University Hospital, Daegu
  - Daejeon Eulji Medical Center, Eulji University, Daejeon
  - Chosun University Hospital, Gwangju
  - Korea University Anam Hospital, Seoul
  - Kangbuk Samsung Hospital, Seoul
  - Yonsei University Health System Severance Hospital, Seoul
  - Kyung Hee University Hospital at Gangdong, Seoul
  - Samsung Medical Center, Seoul
  - Ulsan University Hospital, Ulsan

IPD SHARING:
Plan to Share IPD: Yes
Celltrionpharm makes patient-level, de-identified data sets and associated documents available for all interventional studies after applicable marketing approvals and commercial availability have been received (or program is completely terminated), and an opportunity for the primary publication of the research and final report development has been allowed. To obtain access, researchers must submit a legitimate academic research proposal for adjudication by an independent review panel, who will review the scientific merit of the research and the requestor's qualifications and conflict of interest that can result in potential bias. Once approved, qualified researchers who sign a data sharing agreement are provided access to these data in a secure research environment.